CLINICAL TRIAL: NCT06304584
Title: Rehabilitation of Older High-risk Patients Treated for a Fragility Fracture of the Hip - a Cross-sectoral Study Between Bispebjerg-Frederiksberg Hospital and Frederiksberg Municipality - the HipFracture-Rehab1 Project
Brief Title: Cross-sectoral Rehabilitation of Older High-risk Patients with Hip Fracture
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Frederiksberg Municipality (Unknown)
Responsible Party: Principal Investigator, Morten Tange Kristensen, Professor, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: P-2023-143
Record Dates: First submitted 2024-02-08; First posted 2024-03-12 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Hip Fractures; Rehabilitation; Recovery of Function
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about and monitor the cross-sectoral rehabilitation process in older high-risk patients treated for at fragility fracture of the hip.

The main questions aim to answer:

* how patients are doing up to one year after hip fracture surgery on different outcomes across the continuum of rehabilitation being offered
* what expectations, experiences and satisfaction patients have for the overall rehabilitation process after a hip fracture

Participants age 65 and above with home address in Frederiksberg municipality, living in own home, admitted and treated for at hip fracture at Department of Orthopedic Surgery, Bispebjerg Hospital, will be asked for participation.

DETAILED DESCRIPTION:
In addition to primary and secondary outcome measures some of the patients will be asked to respond to a interviewer-based questionnaire, about their experiences of the rehabilitation offered during their hospital stay and at the temporary municipality-based 24-hour setting / or at home during the first couple of months. Furthermore, they will be interviewed about their expectations for rehabilitation in the municipality at time of discharge from the acute hospital.

ELIGIBILITY:
Inclusion Criteria:

Undergone surgery for hip fracture and admitted to department M1, Bispebjerg-Frederiksberg Hospital

Living in Frederiksberg municipality and being admitted from own home, or a 24 hour temporary setting in the municipality

Exclusion Criteria:

Living permanent in nursing home or is on the way to a permanent nursing home from a 24-hour setting.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be recruited from Bispebjerg Hospital, department M1
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Recovery of pre-fracture function | Recovery of pre-fracture function at 3-4 months post-fracture as primary outcome
  Recovery of function related to the pre-fracture level (re-call last week before fracture) will be assessed with New mobility Score (score 0-9) pre-fracture, at start and end of rehabilitation in municipality, 3-4 month and 1 year post-fracture

SECONDARY OUTCOMES:
Basic mobility | Pre-fracture, at inclusion and discharge from hospital, at start and end of rehabilitation in municipality, 3-4 months and 1 year post-fracture
  Will be measured using Cumulated Ambulation Score (CAS). It describes the patients' independence in three activities (getting in and out of bed, sit-to-stand from a chair, and walking), with each activity assessed on a three-point ordinal scale from 0 to 2, resulting in a total CAS between 0 and 6 (6 is maximum score indicating the patient to be independent in basic mobility).
30 second chair stand test (CST) | At inclusion and discharge from hospital, at start and end of rehabilitation in municipality and 3-4 months post-fracture
  CST test measures how many times a person can stand up from a chair in 30 seconds, without using their arms.
Timed Up & Go test (TUG) | At start and end of rehabilitation in municipality and 3-4 months post-fracture
  TUG test measures the time in seconds it takes a person to stand up from a regular chair with back and armrests, walk 3 meters, turn around, go back to the chair and sit down again
Hip related pain | At inclusion and discharge from hospital, at start and end of rehabilitation in municipality, 3-4 months and 1 year post-fracture
  Will be assessed using the 5-point Verbal Rating Scale (VRS, no pain, slight pain, moderate pain, severe pain, and unbearable pain) during weight-bearing activities
Hand Grip Strength (HGS) | At inclusion at the hospital, at start and end of rehabilitation in municipality and 3-4 months post-fracture
  HGS measures how much strength a person has in their dominant hand. If the dominant hand is injured (e.g. by paralysis or fracture), the test is carried out with the non-dominant hand. Although the measure of HGS assesses the function of one muscle group, it is regarded as an indicator of overall body strength.
Health questionnaire | At pre-fracture (recall) and 3-4 months and 1-year post-fracture
  Will be assessed by the EQ-5D-5L questionnaire. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Physical activity (weekly) | At inclusion (recall of the last few weeks before present hospitalization) and 1-year post-fracture
  Will be assessed using a validated questionnaire from the Swedish National Board of Health and Welfare, providing a total score from 3 to 19. A score ≥11 corresponds to fulfillment of the Word Health Organization's recommendation for weekly physical activity
Physical activity / upright time (time standing and walking) | From inclusion until 9 days post-discharge
  Will be measured using SENS Innovation Aps motion activity measurement system which is a waterproof activity sensor placed laterally on the opposite thigh of the fractured hip.
Frailty | At pre-fracture (recall) and 1-year post-fracture
  Will be assessed using Clinical Frailty Scale (CFS) which is a clinical judgement-based frailty tool. The CFS evaluates specific domains including comorbidity, function., and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Fear of falling | At discharge and 3-4 months and 1-year post-fracture
  Will be assessed with Short-Falls Efficacy Scale, minimum 7 (no concern about falling) to maximum 28 (severe concern about falling). Assesses fear of falling conceptualized as concerns about falling in an 7 item questionnaire.
Comorbidity | At inclusion
  Will be assessed using The American Society of Anesthesiologists (ASA) physical status classification system. The ASA score is a subjective assessment of a patient's overall health that is based on five classes. One means the patients is healthy and fit, and 5 is a moribund patient who is not expected to live 24 hour with or without surgery.
Cognitive status | At inclusion
  Will be assessed using the Short Orientation-Memory Concentration (OMC). It consists of a 6-item patient reported questionnaire and is validated as a measure of cognitive impairment. The score ranges from 0-28 where 0 is equal to normal cognition and 28 is appraised as a severe impairment.
Number of falls | At start and end of rehabilitation in municipality, 3-4 months and 1 year post-fracture
  Place and cause
Residential status / discharge destination | At discharge from hospital and 24-hour rehabilitation setting
  Residential status pre-fracture and discharge destination
Length of stay in acute hospital | From surgery till discharge
  Number of days
Number of weekly exercise sessions with therapist in all settings | At discharge and end of rehabilitation in municipality
  The number of weekly exercise sessions with therapist at hospital, and in the municipality
Number of rehab weeks | At end of rehabilitation in municipality
  In the municipality
Type of training in Municipality | At end of rehabilitation in the Municipality
  Type of rehabilitation with a physiotherapist in Frederiksberg Municipality, at home or individual or team training in the centre, or a mixture of both
Training after discharge from 24-hour setting | At discharge from 24-hour setting
  If the patient has been on a 24-hour setting, is training then continued after discharge
Home care, nurse/other health assistance, times pr week | At pre-fracture, at start and end of rehabilitation in municipality and 3-4 months and 1-year post-fracture
  Assistance with personal care, preparing dinner, grocery shopping, cleaning etc
Data 30 days post-discharge | 30 day post-discharge
  The patient record will be reviewed and it will be recorded if the patient has been readmitted or has died.
Data 3 months post-discharge | 3 month post-discharge
  The patient record will be reviewed and it will be recorded if the patient has been readmitted or has died.
Data 1 year post-discharge | 1 year post-discharge
  The patient record will be reviewed and it will be recorded if the patient has undergone reoperation or has died.

CONTACTS AND LOCATIONS:
Overall Officials: Morten T Kristensen, Professor, Study Chair — Fysio- og Ergoterapien, Bispebjerg-Frederiksberg Hospital
Locations (1):
- Department of Physio- and Occupational Therapy and Othopedic Surgery, University Hospital Bispebjerg and Frederiksberg, Copenhagen, Denmark